CLINICAL TRIAL: NCT05639881
Title: Enhancing Immune Health Literacy and Behavior Among People With Psychiatric Disabilities
Brief Title: Enhancing Immune Health Randomized Controlled Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Institute on Disability, Independent Living, and Rehabilitation Research (U.S. Federal Agency)
Responsible Party: Principal Investigator, Judith A. Cook, Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: STUDY2022-1075
Record Dates: First submitted 2022-11-01; First posted 2022-12-06 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Mental Disorder
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Intervention Model Description: The intervention improves health literacy and self-management skills using a framework comprised of the psychoeducational strategies of explanation, evaluation, and engagement. Over the course of 5 structured sessions, instructors impart immune health information using visual aids. They evaluate what participants already know about immune health to assess how to expand participants' understanding of immunity and health self-management. Instructors engage participants in personally-meaningful activities and goals to improve their immune health literacy and behaviors. For 3 months after class ends, monthly booster sessions are held.
Who Masked: Outcomes Assessor
Masking Description: Research interviewers are blinded to study condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Intervention (Experimental): Subjects receive a brief intervention to improve their immune health literacy and self-management skills.
  Interventions: Behavioral: Enhancing Your Immune Health
- Services as Usual (Active Comparator): Subjects receive routine mental health care.
  Interventions: Behavioral: Enhancing Your Immune Health

INTERVENTIONS:
Behavioral: Enhancing Your Immune Health — In addition to routine mental health care, subjects receive an intervention to improve their immune health literacy and self-management behaviors.

SUMMARY:
This study tests a psychosocial intervention to improve immune health literacy and behaviors among adults with mental illnesses.

DETAILED DESCRIPTION:
This study is testing the efficacy of a brief intervention designed to improve immune health literacy and behaviors among adults with mental illnesses. This psychoeducational intervention supports lifestyle changes, including promotion of immunity-enhancing nutrition and immunity aids, activated intentions to receive needed inoculations and annual health screenings, better sleep, and more effective stress management. Adult clients of collaborating community mental health agencies are randomly assigned to the intervention plus services as usual, versus services as usual alone. They are assessed at baseline, two months post-baseline, and three months later. Multivariable analysis models are used to assess the primary outcome of self-reported immune status.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and older
* Serious mental illness
* Membership in a collaborating community mental health agency
* Access to the Internet
* Able to provide informed consent

Exclusion Criteria:

* Cognitive impairment preventing informed consent
* Unable to communicate in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in Immune Status | study entry (pre-intervention), immediate post-intervention, 3 months post-intervention
  The Immune Status Questionnaire (ISQ) measures self-reported immune status. The questionnaire consists of 7 items measuring indicators of immune health including headache, muscle and joint pain, cough, and sudden high fever. Respondents rate each item using a 5-point Likert scale ranging from "never" to "always or almost always." Responses are coded 0-4 and summed for a total score potentially ranging from 0 to 28 with higher scores indicating a poorer immune status.

SECONDARY OUTCOMES:
Change in Perceived Competence for Health Management | study entry (pre-intervention), immediate post-intervention, 3 months post-intervention
  The Perceived Competence for Health Management scale measures participants' feelings of competence about their ability to manage their immune health. This 4-item scale uses a 7-point Likert response format ranging from "not at all true" to "very true." The minimum value is 4 and the maximum is 28, with higher scores indicating a better outcome.
Change in Coping Mastery | study entry (pre-intervention), immediate post-intervention, 3 months post-intervention
  Change in subjects' sense of personal control over important life outcomes is assessed via 7 items of the Coping Mastery Scale rated along a 4-point Likert scale from "strongly disagree" to "strongly agree." Higher values equal better coping mastery. Minimum=2 and maximum=49.
Change in Health Promoting Lifestyle | study entry (pre-intervention), immediate post-intervention, 3 months post-intervention
  The ability to engage in health promoting behaviors and practices is assessed via self-report on a 26-item Health Promoting Lifestyle Profile II scale that yields a total score and 3 subscales measuring nutrition, physical activity, and emotional and spiritual wellness.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Illinois Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No